CLINICAL TRIAL: NCT00978965
Title: Identification of Patients With High Probability of Not or Poorly Responding to Mycophenolate-mofetil (Cellcept®) or Mycophenolate-natrium (Myfortic®) Therapy
Brief Title: Identification of Patients With High Probability of Poorly Responding to Therapy With Mycophenolic Acid Prodrugs
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Guerkan SENGOELGE, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Other Study IDs: MPASNPVienna
Record Dates: First submitted 2009-09-14; First posted 2009-09-17 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Renal Transplantation
Keywords: kidney transplantation; immunosuppression; single nucleotide polymorphism; IMPDH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Genetic: MPA SNP

INTERVENTIONS:
Genetic: MPA SNP — Functional relevant MPA SNP will be sought in patients DNA isolated from leucocytes

SUMMARY:
This study is designed to define groups of patients (among patients with a heart or kidney graft or a glomerular disease and nephrotic range proteinuria) who would either not profit from a therapy with mycophenolate-mofetil (MMF) or need a higher than conventional dose to respond.

Mainly there are 2 possible explanations for inter-patient differences in responsiveness to MMF therapy:

1. Based on a mutation (in this study single nucleotide polymorphisms-SNPs-) in the inosine monophosphate dehydrogenase 2 (IMPDH 2) transcript as the target enzyme of mycophenolic acid (MPA) pathway, MMF cannot exert its effect.
2. Based on a high enzyme activity of IMPDH 2 a higher MMF dose than in the conventional regimens is needed.

To study the significance of these possible explanations there are 4 objectives in this study:

Objective 1: Since there are no data on SNPs with functional relevance in IMPDH 2 transcript, we will first sequence all 14 exons of this gene in their entirety in 100 gender and age matched healthy individuals.

Objective 2: The functional relevance of a detected SNP will be tested in vitro in a lymphocyte proliferation assay using various MPA concentrations.

Objective 3: These functionally relevant SNPs will be searched in patients with kidney graft in a retrospective as well as prospective manner.

Objective 4: Parallel to the genotyping experiments, IMPDH 2 activity and MPA plasma levels will be measured in all patients recruited in the study prospectively.

An association between these SNPs or various IMPDH 2 activity / MPA plasma levels with MMF responsiveness will be examined.

Objective 5: Strongyloides IgG titers are screened to evaluate the prevalence of helminth carriers in patients with immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with a de novo kidney graft and age >18 and < 75

Exclusion Criteria:

* pregnancy
* panel of antigens reactivity > 40%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a de novo kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2009-10; Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Detection of functionally relevant SNPs in IMPDH 2 gene. | 6 months
The association of detected SNPs in inosine monophosphate dehydrogenase-2 transcript or high IMPDH 2 activity with the lack of response to MPA therapy defined as - number of biopsy proven acute rejections in the first year after transplantation | 12 months per patient

SECONDARY OUTCOMES:
Screening for strongyloides IgG titers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Sengölge, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Medicine III, Division of Nephrology, Vienna, Austria